CLINICAL TRIAL: NCT03500900
Title: Effect of the DPP-4 Inhibitor, Vildagliptin, on Gastric Accommodation and Food Intake in Humans
Brief Title: Vildagliptin on Gastric Accommodation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Vildagliptin
Record Dates: First submitted 2018-01-18; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: gastric accommodation; food intake; gastrointestinal hormones
MeSH Terms: interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vildagliptin (Experimental): DPP-4 inhibitor, acute administration (50 mg.)
  Interventions: Drug: Vildagliptin 50 mg
- Placebo (Placebo Comparator): Placebo treatment, acute administration
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Vildagliptin 50 mg — Acute administration of Vildagliptin, 50 mg.
  Arms: Vildagliptin
Drug: Placebo Oral Tablet — Acute administration of placebo tablet
  Arms: Placebo

SUMMARY:
Dipeptidyl peptidase-4 (DPP-4) inactivates glucagon-like peptide-1 (GLP-1). Whether DPP-4 inhibition affects GLP-1 metabolism in vivo and/or food intake remains unknown.

The aim of this study is to evaluate the effect of vildagliptin (DPP-4 inhibitor) on gastric accommodation and ad libitum food intake in healthy volunteers (HVs).These effects will be evaluated in two randomized, placebo-controlled, single-blinded trials. Each protocol will include ten volunteers.

Protocol 1: Sixty minutes after treatment a nutrient drink (270 kcal) will be intragastrically infused and intragastric pressure (IGP) will be measured for one hour.

Protocol 2: 60 min after treatment the participants consume one nutrient drink (300 kcal). Thirty minutes hereafter, the participant will eat ad libitum from a free-choice buffet for 30 minutes. Blood will be collected at several time points to measure active GLP-1 plasma levels.

ELIGIBILITY:
Inclusion Criteria:

- Aged between 18 to 65 years old

Exclusion Criteria:

* presence of symptoms or a history of gastrointestinal diseases
* diabetes
* drug allergies
* psychological disorders
* major gastrointestinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Change in intragastric pressure measured by high resolution manometry | Until 2 hours after administration of study drug or placebo
  Intragastric pressure will be assessed as a measure for gastric accommodation and gastric motility

SECONDARY OUTCOMES:
Change in subjective gastrointestinal symptom scores measured by visual analogue scale of 100 mm | assessment by questionnaire (100 mm Visual Analogue Scale) every 5 minutes, up to 2 hours after administration
Change in GLP-1 plasma concentrations | Blood samples to assess active GLP-1 plasma levels were collected immediately before medication or placebo administration, 55 minutes, 75 minutes and 120 minutes after medication or placebo administration.
Ad libitum food intake in grams | Buffet was served 1,5 hour after intake of study medication or placebo. Participants had 30 minutes to eat ad libitum until maximal satiation.
  Food items were weighed before and after the buffet to measure food intake in grams.
Ad libitum food intake in kcal | Buffet was served 1,5 hour after intake of study medication or placebo. Participants had 30 minutes to eat ad libitum until maximal satiation.
  Caloric intake of each of the consumed food items was calculated for each subject in a unit of kcal

IPD SHARING:
Plan to Share IPD: No